CLINICAL TRIAL: NCT05358821
Title: A 28-Day Randomized, Placebo-Controlled, Double-Blind, Parallel Groups and Normative Comparison Study to Evaluate the Effect of SAGE-718 on Functioning Capacity in Participants With Huntington's Disease
Brief Title: 28-Day Study of SAGE-718 on Functioning Capacity in Participants With Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 718-CIH-202
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAGE-718 (Experimental): Participants with HD will receive SAGE-718 1.2 milligrams (mg), orally, once daily for up to 28 days.
  Interventions: Drug: SAGE-718
- Placebo (Placebo Comparator): Participants with HD will receive SAGE-718-matching placebo, orally, once daily for up to 28 days.
  Interventions: Drug: Placebo
- Healthy Participants (No Intervention): HP enrolled in this study will not receive any investigational product (IP) (SAGE-718 or placebo).

INTERVENTIONS:
Drug: SAGE-718 — SAGE-718 oral softgel lipid capsules
  Arms: SAGE-718
Drug: Placebo — SAGE-718-matching oral capsules
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the magnitude of the baseline difference between participants with early Huntington's Disease (HD) and healthy participants (HP) with respect to measures of cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

For all

1. Agree to refrain from drugs of abuse for the duration of the study and from alcohol during the 48 hours preceding each study visit.

   Additional criteria for participants with HD only:
2. Be ambulatory, able to travel to the study center, and, judged by the investigator, is likely to be able to continue to travel to the study center to complete study visits for the duration of the study.
3. Have:

   1. Genetically confirmed disease with cytosine, adenine, and guanine (CAG) expansion ≥36.
   2. At screening, Unified Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity (TFC) >6 and <13, suggesting no more than a moderate level of functional impairment.
   3. No features of juvenile HD.
4. CAG-Age-Product (CAP) score >70, as calculated using the CAP formula: Age × (CAG - 30) / 6.49.
5. Score of 15 to 25 (inclusive) on the Montreal Cognitive Assessment (MoCA) at screening, indicating the presence of cognitive impairment.

Additional criteria for HP only:

1. Score ≥26 on the MoCA at screening.
2. Have no known family history of HD; or, have known family history of HD but have genetic test results available that show a normal CAG repeat length for both Huntingtin (HTT) alleles (<36).

Exclusion Criteria:

For All

1. Receive any prohibited medications within 30 days of Screening and during participation in the study
2. Have participated in a previous clinical study of SAGE-718, have previous exposure to gene therapy; or have participated in any HD investigational drug, biologic, or device trial within 180 days, or a non-HD drug, biologic, or device trial within 30 days or 5 half-lives (whichever is longer). (Note: participants with confirmation of enrolment in the placebo arm of these trials would not be excluded.)
3. Is known to be allergic to any of SAGE-718 excipients, including soy lecithin.

Additional criteria for participants with HD only:

1. Had gastric bypass surgery, has a gastric sleeve or lap band, or has had any related procedures that interfere with gastrointestinal transit.
2. Receive any prohibited medications within 30 days of Screening and during participation in the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - Sage Investigational Site, Birmingham, Alabama
  - Sage Investigational Site, Los Alamitos, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Washington D.C., District of Columbia
  - Sage Investigational Site, Boca Raton, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Baltimore, Maryland
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Philadelphia, Pennsylvania
  - Sage Investigational Site, Houston, Texas
- Sage Investigational Site, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 14 investigative sites in the United States and Canada from 26 May 2022 to 10 April 2024.
Pre-assignment Details: A total of 69 adult participants, comprising 29 healthy participants (HP) and 40 participants with Huntington's disease (HD) were enrolled in the study. Participants with HD received either SAGE-718 or placebo. As pre-specified in the protocol, HP enrolled in the study followed the same assessment schedule as participants with HD, but did not receive any investigational product (IP) (SAGE-718 or placebo).
Groups:
- Placebo: Participants with HD received SAGE-718-matching placebo, orally, once daily for up to 28 days.
- SAGE-718: Participants with HD received SAGE-718 1.2 milligrams (mg), orally, once daily for up to 28 days.
- Healthy Participants: HP enrolled in this study did not receive any IP (SAGE-718 or placebo).
Period: Overall Study
Arm/Group | Placebo | SAGE-718 | Healthy Participants
Started | 19 | 21 | 29
Completed | 19 | 20 | 28
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants with HD and all HP who met the eligibility criteria and had at least one baseline assessment of Huntington's disease cognitive assessment Battery (HD-CAB) (participants with HD and HP).
Groups:
- SAGE-718: Participants with HD received SAGE-718 1.2 mg, orally, once daily for up to 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-718 | Healthy Participants | Total
Number analyzed (Participants) | 19 | 21 | 29 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (8.45) | 49.5 (7.44) | 43.5 (11.15) | 47.0 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 14 | 33
  Male | 10 | 11 | 15 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 4 | 9
  Not Hispanic or Latino | 15 | 20 | 25 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Black or African American | 1 | 0 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 18 | 20 | 20 | 58
  Multiple | 0 | 0 | 1 | 1
  Other | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Difference in Huntington's Disease Cognitive Assessment Battery (HD-CAB) Composite Score Between Participants With HD vs HP at Baseline
Description: HD-CAB assesses cognitive function using 6 subtests:Symbol Digit Modalities Test-correctly coded items(0-110); One Touch Stockings of Cambridge(OTS)-mean time to reach correct response(range not defined); Trail Making Test Trail B (TMT-B)-time to complete task(0-240 sec); Hopkins Verbal Learning Test Revised-total correct recall trials(0-48); Paced Tapping Test-reciprocal of standard deviation(SD) of intertap intervals (range not defined); Emotion Recognition Test-negative emotions correctly identified(0-24). Values of OTS & TMT B are multiplied by -1 to represent higher is better direction as other tests. Each of 6 subtests scores was transformed to z-score(range not defined;low negative value represents cognitive impairment), which is calculated by subtracting mean and dividing by SD of HP at baseline. HD-CAB composite=average of 6 z-scores. Negative HD-CAB of HD participants=decline in cognitive function relative to HP. Assessment is relative to reference group(healthy population).
Time Frame: Baseline
Population: FAS included all randomized participants with HD & all HP who met eligibility criteria & had at least 1 baseline assessment of HD-CAB (participants with HD & HP). As primary analysis was to estimate baseline differences between participants with HD & HP in HD-CAB composite score, data from SAGE-718 & placebo arms were combined for analysis. Baseline for HD participants=last non-missing measurement prior to first dose of IP. Baseline for HP=last non-missing measurement on or prior to Day 1.
Measure: Mean (Standard Deviation); unit: Z score
Groups:
- Participants With HD: All participants with HD who were enrolled and randomized into the study to receive either Sage-718 or placebo.
Arm/Group | Participants With HD | Healthy Participants
Number analyzed (Participants) | 40 | 29
Z score | -3.3657 (1.4613) | 0.0000 (0.5673)
Statistical Analysis 1: Comparison: Participants With HD vs Healthy Participants; Test type: Superiority; p < 0.0001, T-test; Mean Difference = 3.3657, 95% CI 2-sided [2.8566 to 3.8749], Standard Error of Mean 0.2539 — Difference was calculated as HP - HD

2. Secondary Outcome: Number of Participants With HD With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Treatment-emergent adverse events are defined as any adverse events with onset on or after the first dose of IP. A serious TEAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death (a life-threatening event), requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, results in a congenital abnormality or birth defect.
Time Frame: Up to Day 42
Population: Safety Set included all participants with HD who were administered IP or HP who met eligibility criteria and was used to describe the safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 19 | 21
Participants
  TEAEs | 6 | 11
  Serious TEAEs | 0 | 0

3. Secondary Outcome: Number of Participants With HD With Clinically Significant Change From Baseline in Vital Sign Measurements
Description: Vital signs including oral temperature, respiratory rate, heart rate (supine and standing), and blood pressures (supine and standing). Number of participants with clinically significant change in vital signs measurements which were deemed clinically significant by the investigator were reported.
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 19 | 21
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With HD With Clinically Significant Change From Baseline in Clinical Laboratory Assessments
Description: Clinical laboratory assessments including hematology, serum chemistry, coagulation, and urinalysis were performed. Number of participants with clinically significant change in laboratory assessments which were deemed clinically significant by the investigator were reported.
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 19 | 21
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 42
Description: Safety Set included all participants with HD who were administered IP or HP who met eligibility criteria and will be used to describe the safety data.
Arm/Group | Placebo | SAGE-718 | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/29
Other Adverse Events (participants affected / at risk) | 6/19 | 7/21 | 4/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | SAGE-718 (N=21) | Healthy Participants (N=29)
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2
Somnolence (Nervous system disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Reflexes abnormal (Nervous system disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT05358821/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT05358821/SAP_001.pdf